CLINICAL TRIAL: NCT03476616
Title: Hypertension thErapy With irBesartan Versus EpleRenone for Obese Patients: A Randomized Clinical Trial
Brief Title: Antihypertensive Pharmacological Therapy With Mineralocorticoid Receptor Antagonists in Obese Hypertensive Patients
Acronym: HEBRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Principal Investigator. Prof. Konstantinos P.Tsioufis, MD, PhD, FESC, FACC, Associate Professor of Cardiology, Head of Hypertension Unit, ESH Excellesh center, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEBRO
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Obesity
Keywords: Hypertension; Obesity; Ambulatory Blood Pressure; Eplerenone; Valsartan; Mineralocorticoid Receptor Antagonists; Angiotensin II Receptor Blockers
MeSH Terms: conditions — Hypertension; Obesity | interventions — Eplerenone; Valsartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eplerenone (-based therapy) arm (Active Comparator): Obese pts with hypertension, starting treatment with eplerenone 25mg twice daily (BD). ABPM wil be scheduled at wks 8, 16 and 24.
  At wk 8 if mean ABPM < 130/80mm Hg will continue to monotherapy with eplerenone. If not controlled (mean ABPM > 130/80mm Hg) at wk8, amlodipine 5mg OD will be added.
  At wk 16 if mean ABPM < 130/80mm Hg will continue to monotherapy with eplerenone, or dual therapy with eplerenone and amlodipine. If not controlled (mean ABPM > 130/80mm Hg) at wk16, indapamide 1,5mg OD will be added. All patients will be followed up for 24 weeks.
  Interventions: Drug: Eplerenone (-based therapy) arm
- Irbesartan (-based therapy) arm (Active Comparator): Obese pts with hypertension, starting treatment with irbesartan 150mg once daily (OD). ABPM wil be scheduled at wks 8, 16 and 24.
  At wk 8 if mean ABPM < 130/80mm Hg will continue to monotherapy with irbesartan. If not controlled (mean ABPM > 130/80mm Hg) at wk8, amlodipine 5mg OD will be added.
  At wk 16 if mean ABPM < 130/80mm Hg will continue to monotherapy with irbesartan, or dual therapy with irbesartan and amlodipine. If not controlled (mean ABPM > 130/80mm Hg) at wk16, indapamide 1,5mg OD will be added. All patients will be followed up for 24 weeks.
  Interventions: Drug: Valsartan (-based therapy) arm

INTERVENTIONS:
Drug: Eplerenone (-based therapy) arm — At randomization, pts meeting inclusion/exclusion criteria will be randomized (1:1) to either eplerenone (E) 25mg bd or valsartan (V) 160mg od for 8 wks. At 8, 16 and 24 wks, pts at both arms will be evaluated with ABPM primary, as well as home and office BP measurements. At wk 8, pts with controlled hypertension (mean ABPM <130/80mmHg), will continue in monotherapy with eplerenone or valsartan and pts with uncontrolled hypertension (mean ABPM ≥130/80mmHg) will continue with the addition of amlodipine (C) 10mg od. At wk 16, pts achieving BP control will continue in either monotherapy (E), (V) or dual therapy (E+C), (V+C). However, in pts not achieving ABPM target, a third drug, will be added [indapamide (D) 1.25 mg od]. All groups at both arms will be evaluated at 24 wks by ABPM.
  Arms: Eplerenone (-based therapy) arm
Drug: Valsartan (-based therapy) arm — At randomization, pts meeting inclusion/exclusion criteria will be randomized (1:1) to either eplerenone (E) 25mg bd or valsartan (V) 160mg od for 8 wks. At 8, 16 and 24 wks, pts at both arms will be evaluated with ABPM primary, as well as home and office BP measurements. At wk 8, pts with controlled hypertension (mean ABPM <130/80mmHg), will continue in monotherapy with eplerenone or valsartan and pts with uncontrolled hypertension (mean ABPM ≥130/80mmHg) will continue with the addition of amlodipine (C) 10mg od. At wk 16, pts achieving BP control will continue in either monotherapy (E), (V) or dual therapy (E+C), (V+C). However, in pts not achieving ABPM target, a third drug, will be added [indapamide (D) 1.25 mg od]. All groups at both arms will be evaluated at 24 wks by ABPM.
  Arms: Irbesartan (-based therapy) arm

SUMMARY:
Obesity is a complex metabolic state at which many pathophysiological pathways seem to interfere, like imbalance of autonomic nervous system, as well as renin-angiotensin-aldosterone system (RAAS) activation. Latest studies have shown that the increase of peripheral fat in obese patients, alongside with the increase of P-450 aromatase leads to hyper-aldosteronism, which results to increased sodium intake and rise of blood pressure. The present study aims to investigate the potential superiority of an aldosterone antagonist based therapy (eplerenone) over the renin-angiotensin antagonists (ARBs) (valsartan) based therapy in hypertensive obese patients regarding reduction of blood pressure (office, home and ambulatory) over a 24-week period.

DETAILED DESCRIPTION:
The present study plans to enroll obese patients (BMI= 30-40 kg/m2) of 30-75 years of age, with untreated or never-treated essential hypertension to either eplerenone-based or irbesartan-based therapy Patients visiting hypertension center(s), eligible to participate in the study and meeting study's inclusion criteria, will at first thoroughly be informed of study's protocol rationale, including scheduled follow-up visits. There will be a period of 2-4 weeks, at which medical history will be taken, as well as somatometrics, including height, weight, BMI and waist circumference. Moreover, a thorough clinical examination will take place, including office blood pressure, ECG, heart-echo, renal ultrasound, blood and urine ultrasound. All women of gestational age should have pregnancy test.

At randomization visit, patients still meeting inclusion/exclusion criteria will be randomized (1:1) to either eplerenone (E) 25mg bd or irbesartan (I) 150mg od for 8 weeks. At 8, 16 and 24 weeks, patients at both arms will be evaluated with ambulatory BP measurements primary, as well as home and office BP measurements. At week 8, patients with controlled blood pressure (mean ambulatory blood pressure measurement (ABPM) <130/80mmHg), will continue in monotherapy with eplerenone or irbesartan and patients with uncontrolled hypertension (mean 24-h ambulatory≥130/80mmHg) will continue with the addition of calcium-channel blocker, amlodipine (C) 5 mg od. At week 16, patients achieving BP control will continue in either monotherapy (E), (I) or dual therapy (E+C), (I+C). However, in patients not achieving blood pressure target, a third drug, thiazide-like-diuretic will be added [indapamide (D) 1.25 mg od]. All groups at both arms will be finally evaluated at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 30-75 years of age
2. Written consent
3. Untreated or never-treated arterial hypertension with office systolic blood pressure of 140-180 mmHg and/or diastolic blood pressure of 90-120 mmHg, confirmed by 24-hour ambulatory blood pressure measurements of mean ambulatory systolic blood pressure over 130 mmHg and/or mean ambulatory diastolic blood pressure over 80 mmHg
4. Obesity, confirmed estimated by Body Mass Index (BMI) of 30-40 kg/m2

Exclusion Criteria

1. Age <30 or >75
2. Inability to give informed consent
3. Participation in a clinical study involving an investigational drug or device within 4 weeks of screening
4. Secondary hypertension
5. Recent (<6 months) cardiovascular event requiring hospitalization (eg. myocardial infarction or stroke)
6. Type 1 diabetes
7. Chronic kidney disease assessed by Estimated Glomerular Filtration Rate (eGFR) <45 mL/min
8. Bilateral renal arteries stenosis
9. Addison's disease
10. Hemodynamically significant valvular heart disease
11. Plasma potassium outside of normal range on two successive measurements during screening
12. Pregnancy, planning to conceive or women of childbearing potential, that is, not using effective contraception
13. Scheduled surgery or cardiovascular surgery over the next 6 months
14. Absolute contra-indication to study drugs (eg. asthma) or previous intolerance of trial therapy
15. History of sustained atrial fibrillation
16. Requirement for study drug for reason other than to treat hypertension, (eg, β-blockers for angina or aldosterone antagonists for heart failure)
17. Neoplasm under treatment (radiotherapy / chemotherapy / immunotherapy)
18. Any concomitant condition that, in the opinion of the investigator, may adversely affect the safety and/or efficacy of the study drug or
19. severely limit that patients' life-span or ability to complete the study (eg, alcohol or drug abuse, disabling or terminal illness, mental
20. disorders)
21. Contemporary systemic disease with life expectancy shorter than the end of the study
22. Treatment with any of the following medications:

    * Oral corticosteroids within 3 months of screening. Treatment with systemic corticosteroids is also prohibited during study participation
    * Chronic stable use, or unstable use of NSAIDs (other than low dose aspirin) is prohibited. Chronic use is defined as >3 consecutive or non-consecutive days of treatment per week. In addition, intermittent use of NSAIDs is strongly discouraged throughout the study and NSAIDs if required, must not be used for more than a total of 2 days. For those requiring analgesics during the study, paracetamol is recommended.
    * The use of short-acting nitrates (eg, sublingual nitroglycerin) is permitted.
    * The use of sympathomimetic decongestants is permitted, however, not within 1 day prior to any study visit/BP assessment
    * The use of theophylline is permitted but the dose must be stable for at least 4 weeks prior to screening and throughout the study;
    * The use of phosphodiesterase type V inhibitors is permitted; however, study participants must refrain from taking these medications for at least 1 day prior to screening or any subsequent study visits
    * The use of α-blockers is not permitted, with the exception of alfuzosin and tamsulosin for prostatic symptoms

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in change of ABPM from baseline, in the eplerenone arm versus the irbesartan arm as monotherapy at 8 weeks, as combined dual treatment with amlodipine at 16 weeks and as combined triple treatment with amlodipine and indapamide at 24 weeks. | 8, 16 and 24 weeks
  Ambulatory blood pressure measurements (metric unit: mmHg) at baseline and 8,16 and 24 weeks and evaluation of the difference of mean ambulatory systolic and diastolic blood pressure measurements between baseline and each time frame in all participants

SECONDARY OUTCOMES:
Difference in change of office BP from baseline, in the eplerenone arm versus the valsartan arm as monotherapy at 8 weeks, as combined dual treatment with amlodipine at 16 weeks and as combined triple treatment with amlodipine and indapamide at 24 weeks. | 8, 16 and 24 weeks
  Office blood pressure measurements (metric unit: mmHg) at baseline and 8,16 and 24 weeks and evaluation of the difference of office systolic and diastolic blood pressure measurements between baseline and each time frame in all participants

OTHER OUTCOMES:
Difference in frequency of controlled hypertension (mean ABPM < 130/80 mm Hg) between the study arms at 8, 16 and 24 weeks. | 8, 16 and 24 weeks
  Ambulatory blood pressure monitoring (metric unit: mmHg) at baseline and 8,16 and 24 weeks and evaluation of the difference of mean ambulatory systolic and diastolic blood pressure measurements between baseline and each time frame in all participants

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos P Tsioufis, Ass. Prof., Principal Investigator — Hypertension Unit, First Cardiology Clinic, Hippocration General Hospital, University of Athens, Greece
Locations (1):
- Hypertension Unit, First Cardiology Clinic, Hippocration General Hospital, University of Athens, Athens, Greece, Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsioufis C, Tsiachris D, Dimitriadis K, Thomopoulos C, Syrseloudis D, Andrikou E, Chatzis D, Taxiarchou E, Selima M, Mazaraki A, Chararis G, Tolis P, Gennadi A, Andrikou I, Stefanadi E, Fragoulis V, Tzamou V, Panagiotakos D, Tousoulis D, Stefanadis C. Leontio Lyceum ALbuminuria (3L Study) epidemiological study: aims, design and preliminary findings. Hellenic J Cardiol. 2009 Nov-Dec;50(6):476-83. PMID 19942561
- [Background] Schlaich MP, Grassi G, Lambert GW, Straznicky N, Esler MD, Dixon J, Lambert EA, Redon J, Narkiewicz K, Jordan J; European Society of Hypertension Working Group on Obesity; Australian and New Zealand Obesity Society. European Society of Hypertension Working Group on Obesity Obesity-induced hypertension and target organ damage: current knowledge and future directions. J Hypertens. 2009 Feb;27(2):207-11. doi: 10.1097/HJH.0b013e32831dafaf. No abstract available. PMID 19155773
- [Background] Dimitriadis K, Tsioufis C, Mazaraki A, Liatakis I, Koutra E, Kordalis A, Kasiakogias A, Flessas D, Tentolouris N, Tousoulis D. Waist circumference compared with other obesity parameters as determinants of coronary artery disease in essential hypertension: a 6-year follow-up study. Hypertens Res. 2016 Jun;39(6):475-9. doi: 10.1038/hr.2016.8. Epub 2016 Feb 11. PMID 26865004
- [Background] Tsioufis CP, Tsiachris DL, Selima MN, Dimitriadis KS, Thomopoulos CG, Tsiliggiris DC, Gennadi AS, Syrseloudis DC, Stefanadi ES, Toutouzas KP, Kallikazaros IE, Stefanadis CI. Impact of waist circumference on cardiac phenotype in hypertensives according to gender. Obesity (Silver Spring). 2009 Jan;17(1):177-82. doi: 10.1038/oby.2008.462. Epub 2008 Oct 23. PMID 18948974
- [Background] Jordan J, Yumuk V, Schlaich M, Nilsson PM, Zahorska-Markiewicz B, Grassi G, Schmieder RE, Engeli S, Finer N. Joint statement of the European Association for the Study of Obesity and the European Society of Hypertension: obesity and difficult to treat arterial hypertension. J Hypertens. 2012 Jun;30(6):1047-55. doi: 10.1097/HJH.0b013e3283537347. PMID 22573071
- [Background] Badimon L, Bugiardini R, Cenko E, Cubedo J, Dorobantu M, Duncker DJ, Estruch R, Milicic D, Tousoulis D, Vasiljevic Z, Vilahur G, de Wit C, Koller A. Position paper of the European Society of Cardiology-working group of coronary pathophysiology and microcirculation: obesity and heart disease. Eur Heart J. 2017 Jul 1;38(25):1951-1958. doi: 10.1093/eurheartj/ehx181. No abstract available. PMID 28873951
- [Background] Doll S, Paccaud F, Bovet P, Burnier M, Wietlisbach V. Body mass index, abdominal adiposity and blood pressure: consistency of their association across developing and developed countries. Int J Obes Relat Metab Disord. 2002 Jan;26(1):48-57. doi: 10.1038/sj.ijo.0801854. PMID 11791146
- [Background] Mancia G, Bombelli M, Corrao G, Facchetti R, Madotto F, Giannattasio C, Trevano FQ, Grassi G, Zanchetti A, Sega R. Metabolic syndrome in the Pressioni Arteriose Monitorate E Loro Associazioni (PAMELA) study: daily life blood pressure, cardiac damage, and prognosis. Hypertension. 2007 Jan;49(1):40-7. doi: 10.1161/01.HYP.0000251933.22091.24. Epub 2006 Nov 27. PMID 17130308
- [Background] Tsioufis C, Tatsis I, Thomopoulos C, Wilcox C, Palm F, Kordalis A, Katsiki N, Papademetriou V, Stefanadis C. Effects of hypertension, diabetes mellitus, obesity and other factors on kidney haemodynamics. Curr Vasc Pharmacol. 2014 May;12(3):537-48. doi: 10.2174/157016111203140518173700. PMID 23305375
- [Background] Cushman WC, Ford CE, Cutler JA, Margolis KL, Davis BR, Grimm RH, Black HR, Hamilton BP, Holland J, Nwachuku C, Papademetriou V, Probstfield J, Wright JT Jr, Alderman MH, Weiss RJ, Piller L, Bettencourt J, Walsh SM; ALLHAT Collaborative Research Group. Success and predictors of blood pressure control in diverse North American settings: the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). J Clin Hypertens (Greenwich). 2002 Nov-Dec;4(6):393-404. doi: 10.1111/j.1524-6175.2002.02045.x. PMID 12461301
- [Background] Hall JE, Brands MW, Dixon WN, Smith MJ Jr. Obesity-induced hypertension. Renal function and systemic hemodynamics. Hypertension. 1993 Sep;22(3):292-9. doi: 10.1161/01.hyp.22.3.292. PMID 8349321
- [Background] Engeli S, Negrel R, Sharma AM. Physiology and pathophysiology of the adipose tissue renin-angiotensin system. Hypertension. 2000 Jun;35(6):1270-7. doi: 10.1161/01.hyp.35.6.1270. PMID 10856276
- [Background] de Paula RB, da Silva AA, Hall JE. Aldosterone antagonism attenuates obesity-induced hypertension and glomerular hyperfiltration. Hypertension. 2004 Jan;43(1):41-7. doi: 10.1161/01.HYP.0000105624.68174.00. Epub 2003 Nov 24. PMID 14638627
- [Background] Garg R, Kneen L, Williams GH, Adler GK. Effect of mineralocorticoid receptor antagonist on insulin resistance and endothelial function in obese subjects. Diabetes Obes Metab. 2014 Mar;16(3):268-72. doi: 10.1111/dom.12224. Epub 2013 Oct 31. PMID 24125483
- [Background] de Souza F, Muxfeldt E, Fiszman R, Salles G. Efficacy of spironolactone therapy in patients with true resistant hypertension. Hypertension. 2010 Jan;55(1):147-52. doi: 10.1161/HYPERTENSIONAHA.109.140988. Epub 2009 Oct 26. PMID 19858405
- [Background] Vaclavik J, Sedlak R, Jarkovsky J, Kocianova E, Taborsky M. Effect of spironolactone in resistant arterial hypertension: a randomized, double-blind, placebo-controlled trial (ASPIRANT-EXT). Medicine (Baltimore). 2014 Dec;93(27):e162. doi: 10.1097/MD.0000000000000162. PMID 25501057
- [Background] Williams B, MacDonald TM, Morant S, Webb DJ, Sever P, McInnes G, Ford I, Cruickshank JK, Caulfield MJ, Salsbury J, Mackenzie I, Padmanabhan S, Brown MJ; British Hypertension Society's PATHWAY Studies Group. Spironolactone versus placebo, bisoprolol, and doxazosin to determine the optimal treatment for drug-resistant hypertension (PATHWAY-2): a randomised, double-blind, crossover trial. Lancet. 2015 Nov 21;386(10008):2059-2068. doi: 10.1016/S0140-6736(15)00257-3. Epub 2015 Sep 20. PMID 26414968
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- See also: PROTOCOL OF THE HYPERTENSION THERAPY WITH IRBESARTAN VERSUS EPLERENONE FOR OBESE HYPERTENSIVE PATIENTS (HEBRO) — https://journals.lww.com/jhypertension/abstract/2019/07001/protocol_of_the_hypertension_therapy_with.646.aspx?casa_token=9AEQ4r6H7jQAAAAA:Pe3rRLJQwJgmcd4BQ8j-bGfYuwh5IDkopKUOC2b7j7_dM8vuYZNAqsIH0qqnmmmv2xPIs3XPprKXAwH9-A3PfhPCHn9z8g
- See also: EPLERENONE VS IRBESARTAN AS FIRST LINE THERAPY IN OBESE HYPERTENSIVE PATIENTS: BASELINE CHARACTERISTICS — https://journals.lww.com/jhypertension/abstract/2023/06003/eplerenone_vs_irbesartan_as_first_line_therapy_in.795.aspx?casa_token=4ug7-a4qsb8AAAAA:2oxBy6ImKeOZYXnrjuJ5ClqJCGER4M4FKckBjFfyjyHAcd26smHfk0azK1Pkc2SGiH59FnzCS_jLYBfuUvlwBGwSD_MLnQ